CLINICAL TRIAL: NCT01612468
Title: Liraglutide in Type 1 Diabetes. A Randomised, Double-blind, Placebo Controlled Study of the Effect of Liraglutide as an Additional Treatment to Insulin on HbA1c, Body Weight and Hypoglycaemia in Poorly Regulated Type 1 Diabetes Patients
Brief Title: Liraglutide in Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Lise Tarnow, professor chief physician, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Lira1
Record Dates: First submitted 2012-05-11; First posted 2012-06-05 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus, Type 1; Overweight
Keywords: Diabetes; Liraglutide; Hypoglycaemia; Hyperglycaemia; CIMT; PWV; Food preference; Blood pressure
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Overweight; Diabetes Mellitus; Hypoglycemia; Hyperglycemia; Food Preferences | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental)
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — 1.8 mg/day subcutaneous
  Other Names: Victoza
  Arms: Liraglutide
Drug: Placebo — 1.8 mg/day subcutaneous
  Arms: Placebo

SUMMARY:
A randomised, double-blind, placebo controlled study of the effect of liraglutide as an additional treatment to insulin on HbA1c, body weight and hypoglycaemia in poorly regulated type 1 diabetes patients.

Background: Treatment with glucagon-like peptid 1 (GLP-1) agonists liraglutide and exanatide leads to weight loss and decrease in haemoglobin A1c in oral anti diabetic treated type 2 diabetes patients.

It is estimated that 40-50 % of type 1 diabetes patients in the US suffers from overweight or poor glycaemic control (HbA1c > 8 %).

Small studies, not placebo controlled, reports effects of adding liraglutide to a group of well regulated (HbA1c < 7.5 %) normal to overweight insulin treated type 1 diabetes patients for 24 weeks. A decrease in HbA1c, weight, insulin doses and glycaemic excursions measured by continuous glucose monitoring was seen.

Primary objective:To investigate the effect of liraglutide 1.8 mg once daily compared to placebo for 24 weeks on change in HbA1c in patients with type 1 diabetes as an add-on therapy to insulin. Secondary objectives:To investigate the effect of liraglutide as an add-on therapy to insulin compared to placebo on change in:Weight, insulin dose,hypoglycaemic events, CGM, BMI, body composition, quality of life, treatment satisfaction,food preferences, meal test, CIMT, PWV and 24 hour blood pressure.

DETAILED DESCRIPTION:
A randomised, double-blind, placebo controlled study of the effect of liraglutide as an additional treatment to insulin on HbA1c, body weight and hypoglycaemia in poorly regulated type 1 diabetes patients.

Background Treatment with glucagon-like peptid 1 (GLP-1) agonists liraglutide and exenatide leads to weight loss and decrease in haemoglobin A1c (HbA1c) in oral anti diabetic treated type 2 diabetes patients. Smaller studies have shown similar effects in insulin treated type 2 diabetes patients, with no increased risk of hypoglycaemia.

It is estimated that 40-50 % of type 1 diabetes patients in the US suffers from overweight or poor glycaemic control (HbA1c > 8 %). At present treatment of type 1 diabetes solely consists of insulin injections.

A recent study reports effects of adding liraglutide to a group of well regulated (HbA1c < 7.5 %) normal to overweight insulin treated type 1 diabetes patients for 24 weeks. A decrease in HbA1c, weight, insulin doses and glycaemic excursions measured by continuous glucose monitoring was seen. The study was not placebo controlled.

The available literature suggests that GLP-1 agonists reduce insulin dose and weight in well regulated type 1 diabetes patients, who are normal- to overweight. To our knowledge, no study has addressed whether liraglutide will improve HbA1c and reduce bodyweight in overweight and poorly regulated type 1 diabetes patients.

At present the most efficient way to reduce HbA1c is to use insulin pump therapy, and most studies suggest that this will decreased HbA1c by approximately 0.5 %. Insulin pump therapy is however only an option in very compliant patients. In most clinics treating type 1 diabetes 40-50 % of patients will have HbA1c > 8 % and many of these patients will, due to insufficient compliance, not be candidates for an insulin pump.

At Steno Diabetes Center approximately 3000 well characterized type 1 diabetes patients is followed in the outpatient clinic, and 40-50 % of these have HbA1c > 8.0 %. If liraglutide given once daily results in a reduction of HbA1c of 0.5 % it will probably be a very cost-effective additional therapy for type 1 diabetes patients in insufficient metabolic control.

Several studies have shown that liraglutide lowers systolic blood pressure. Dysregulation increases the risk of microvascular complications in type 1 diabetes of which microalbuminuria results in a need for treatment with antihypertensive medication. Overweight increases the risk of hypertension and arteriosclerosis and thereby cardiovascular diseases. Carotis intima media thickness is a validated estimate for future cardiovascular disease and pulse wave velocity is a measure of arterial stiffness. We perform 24 hour blood pressure measurements to document possible effects of liraglutide on blood pressure and CIMT and PWV to investigate the effect of liraglutide on cardiovascular disease and arteriosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes according to WHO criteria ≥ 1 year
* Age ≥ 18 years
* BMI > 25 kg/m2
* HbA1c > 8.0 % at visit 0

Exclusion Criteria:

* Insulin pump treatment
* Hypoglycaemia unawareness (unability to register low blood glucose)
* Diabetic gastroparesis
* Compromised kidney function (eGFR < 60 ml/min/1,73m2), dialysis or kidney transplantation at visit 0
* Liver disease with elevated plasma alanine aminotransferase (ALT) > three times the upper limit of normal (measured at visit 0 with the possibility of one repeat analysis within a week, and the last measured value as being conclusive)
* Acute or chronic pancreatitis
* Inflammatory bowel disease
* Cancer unless in complete remission for > 5 years
* History of thyroid adenoma or carcinoma
* Other concomitant disease or treatment that according to the investigator's assessment makes the patient unsuitable for study participation
* Alcohol/drug abuse
* Fertile women not using contraceptives
* Pregnant or nursing women
* Known or suspected hypersensitivity to trial product or related products
* Receipt of an investigational drug within 30 days prior to visit 0
* Simultaneous participation in any other clinical intervention trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 24 week
  To investigate the effect of liraglutide 1.8 mg once daily compared to placebo for 24 weeks on change in HbA1c in patients with type 1 diabetes as an adjunctive therapy to insulin treatment.

SECONDARY OUTCOMES:
Body weight | 24 weeks
  To investigate the effect of liraglutide 1.8 mg once daily compared to placebo for 24 weeks on change in weight, BMI and body composition
Cardiovascular | 24 weeks
  To investigate the effect of liraglutide 1.8 mg once daily compared to placebo for 24 weeks on change in carotis intima media thickness, pulse wave velocity, 24 hour blood pressure
Standardised liquid meal test | 24 weeks
  To investigate the effect of liraglutide 1.8 mg once daily compared to placebo for 24 weeks on change in postprandial glucagon levels, glycaemic excursion, gastric emptying, VAS score for appetite and food preference
Glycaemic excursions | 24 weeks
  To investigate the effect of liraglutide 1.8 mg once daily compared to placebo for 24 weeks on change in insulin dose, hypoglycaemic events and glycaemic excursions (time spent in hypo- and hyperglycaemia as measured by CGM)
Quality of life | 24 weeks
  To investigate the effect of liraglutide 1.8 mg once daily compared to placebo for 24 weeks on change in quality of life and treatment satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Henrik U Andersen, DMSc, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Dejgaard TF, Frandsen CS, Hansen TS, Almdal T, Urhammer S, Pedersen-Bjergaard U, Jensen T, Jensen AK, Holst JJ, Tarnow L, Knop FK, Madsbad S, Andersen HU. Efficacy and safety of liraglutide for overweight adult patients with type 1 diabetes and insufficient glycaemic control (Lira-1): a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2016 Mar;4(3):221-232. doi: 10.1016/S2213-8587(15)00436-2. Epub 2015 Dec 3. PMID 26656289
- [Derived] Dejgaard TF, Knop FK, Tarnow L, Frandsen CS, Hansen TS, Almdal T, Holst JJ, Madsbad S, Andersen HU. Efficacy and safety of the glucagon-like peptide-1 receptor agonist liraglutide added to insulin therapy in poorly regulated patients with type 1 diabetes--a protocol for a randomised, double-blind, placebo-controlled study: the Lira-1 study. BMJ Open. 2015 Apr 2;5(4):e007791. doi: 10.1136/bmjopen-2015-007791. PMID 25838513